CLINICAL TRIAL: NCT06136624
Title: A Phase 3 Randomized, Open-label Study of MK-5684 Versus Alternative Abiraterone Acetate or Enzalutamide in Participants With Metastatic Castration-resistant Prostate Cancer (mCRPC) Previously Treated With Next-generation Hormonal Agent (NHA) and Taxane-based Chemotherapy (OMAHA-003)
Brief Title: Study of Opevesostat (MK-5684) Versus Alternative NHA in mCRPC (MK-5684-003)
Acronym: OMAHA-003
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5684-003; 2023-504899-25-00 (Other: EU CT); MK-5684-003 (Other: MSD); jRCT2031240029 (Registry Identifier: Japan Registry of Clinical Trials (jRCT)); U1111-1287-5304 (Registry Identifier: UTN)
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer Metastatic
MeSH Terms: interventions — Abiraterone Acetate; enzalutamide; Hydrocortisone; fludrocortisone acetate; Prednisone; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Opevesostat (Experimental): Participants receive opevesostat 5 mg by oral tablets twice daily (bid) plus dexamethasone 1.5 mg by oral tablets once daily (qd) and 0.1 mg fludrocortisone acetate by oral tablet qd until progression. Hydrocortisone 100 mg (oral or intramuscular [IM]) dose will also be provided to participants for use as rescue medication.
  Interventions: Drug: Opevesostat; Drug: Hydrocortisone; Drug: Fludrocortisone acetate; Drug: Dexamethasone
- Abiraterone Acetate or Enzalutamide (Active Comparator): Participants receive abiraterone 1000 mg qd by oral tablets plus prednisone 5 mg bid by oral tablets or enzalutamide 160 mg qd by oral tablets.
  Interventions: Drug: Abiraterone acetate; Drug: Enzalutamide; Drug: Prednisone

INTERVENTIONS:
Drug: Opevesostat — Administered orally
  Other Names: MK-5684
  Arms: Opevesostat
Drug: Abiraterone acetate — Administered orally
  Other Names: ZYTIGA; YONSA
  Arms: Abiraterone Acetate or Enzalutamide
Drug: Enzalutamide — Administered orally
  Other Names: XTANDI
  Arms: Abiraterone Acetate or Enzalutamide
Drug: Hydrocortisone — Administered orally or IM as a rescue medication
  Arms: Opevesostat
Drug: Fludrocortisone acetate — Administered orally
  Arms: Opevesostat
Drug: Prednisone — Administered orally
  Arms: Abiraterone Acetate or Enzalutamide
Drug: Dexamethasone — Administered orally as rescue medication
  Arms: Opevesostat

SUMMARY:
This is a phase 3, randomized, open-label study of opevesostat compared to alternative abiraterone acetate or enzalutamide in participants with metastatic castration-resistant prostate cancer (mCRPC) with respect to overall survival (OS) in participants with mCRPC previously treated with next-generation hormonal agent (NHA) and taxane-based chemotherapy. It is hypothesized that opevesostat is superior with respect to OS in androgen receptor ligand binding domain (AR LBD) mutation-negative and -positive participants.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically- or cytologically-confirmed adenocarcinoma of the prostate without small cell histology.
* Has prostate cancer progression while on androgen deprivation therapy (or post bilateral orchiectomy) within 6 months before Screening
* Has current evidence of distant metastatic disease (M1 disease) documented by either bone lesions on bone scan and/or soft tissue disease by computed tomography/magnetic resonance imaging (CT/MRI).
* Has disease that progressed during or after treatment with 1 novel hormonal agent (NHA)
* Has received 1 but no more than 2 taxane-based chemotherapy regimens for metastatic castration-resistant prostate cancer (mCRPC) and has had progressive disease (PD) during or after treatment
* Has ongoing androgen deprivation with serum testosterone <50 ng/dL (<1.7 nM)
* Has provided tumor tissue from a fresh core or excisional biopsy from soft tissue not previously irradiated
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 assessed within 7 days of randomization
* Has had prior treatment with PARPi or were deemed ineligible to receive treatment by the investigator or have refused PARPi treatment
* Has received prior 177Lu-PSMA-617 or were deemed ineligible to receive 177Lu-PSMA-617 treatment by the investigator or refused 177Lu-PSMA-617 treatment
* Participants who have not received cabazitaxel can be enrolled if they are ineligible for cabazitaxel treatment as determined by the investigator or have refused treatment
* If participant received first generation anti-androgen therapy before screening, the participant has evidence of disease progression >4 weeks since the last flutamide treatment and >6 weeks since the last bicalutamide or nilutamide treatment
* Participants receiving bone resorptive therapy (including, but not limited to, bisphosphonate or denosumab) must have been on stable doses for ≥ 4 weeks before the date of randomization
* Participants with human immunodeficiency virus (HIV) infection must have well controlled HIV on antiretroviral therapy (ART)
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load before randomization
* Participants with history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at Screening.
* Participants who can produce sperm must agree to the following during the study treatment period and for at least 7 days after the last dose of opevesostat, for at least 30 days after the last dose of abiraterone acetate, and for at least 3 months after the last dose of enzalutamide: EITHER be abstinent OR must agree to use male condom

Exclusion Criteria:

* Has a gastrointestinal disorder that might affect absorption
* Has a history of pituitary dysfunction
* Has poorly controlled diabetes mellitus
* Has clinically significant abnormal serum potassium or sodium level
* Has a history of active or unstable cardio/cerebro-vascular disease, including thromboembolic events
* Has a history of seizure within 6 months of providing documented informed consent or any condition that may predispose to seizures within 12 months before the date of randomization
* Has a history of clinically significant ventricular arrhythmias
* Has received an anticancer monoclonal antibody (mAb) within 4 weeks before the date of randomization, or has not recovered from adverse events (AEs) due to mAbs administered more than 4 weeks before the date of randomization
* Has undergone major surgery, including local prostate intervention (except prostate biopsy), within 28 days before the date of randomization, and has not recovered from the toxicities and/or complications
* Participants who have not adequately recovered from major surgery or have ongoing surgical complications
* Has used herbal or medicinal products that may have hormonal anti-prostate cancer activity and/or are known to decrease prostate-specific Antigen (PSA) (eg, saw palmetto, megesterol acetate, citrus pectin polysaccharide) within 4 weeks before the date of randomization
* Has received radium-223 or lutetium-177 within 4 weeks before the date of randomization, or has not recovered to Grade ≤1 or baseline from AEs due to radium-223 or lutetium-177 administered more than 4 weeks before the date of randomization
* Has received treatment with 5-αreductase inhibitors (eg, finasteride or dutasteride), estrogens, or cyproterone within 4 weeks before the date of randomization
* Has received colony-stimulating factors within 28 days before the date of randomization
* Has received a whole blood transfusion in the last 120 days before the date of randomization. Packed red blood cells and platelet transfusions are acceptable if not given within 28 days of the date of randomization
* Has received prior targeted small molecule therapy or NHA treatment within 4 weeks before the first dose of study intervention as follows: enzalutamide or apalutamide within 3 weeks or abiraterone acetate + prednisone or darolutamide within 2 weeks
* Has a "superscan" bone scan
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior the first dose of study medication
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has an active infection requiring systemic therapy
* Has concurrent active HBV or known active HCV infection
* Has a history of long QTc syndrome
* Has any of the following at Screening Visit: hypotension (systolic BP <110 mm Hg) or uncontrolled hypertension (systolic BP ≥160 mm Hg or diastolic BP ≥90 mm Hg, in 2 out of 3 recordings with optimized antihypertensive therapy)
* Is unable to swallow capsules/tablets
* Is currently being treated with cytochrome 450-inducing antiepileptic drugs for seizures
* Participants on an unstable dose of thyroid hormone therapy within 6 months before the start of the study intervention
* Received prior systemic anticancer therapy including investigational agents within 4 weeks before the first dose of study intervention
* Received prior radiotherapy within 2 weeks of start of study intervention, or radiation-related toxicities, requiring corticosteroids
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Systemic use of the following medications within 2 weeks before the first dose of study intervention: strong CYP3A4 inducers (eg, avasimibe, carbamazepine, lumacaftor, phenobarbital, rifampicin, rifapentine, or St John's Wort); P-gp inhibitors (eg, erythromycin, clarithromycin, rifampicin, ketoconazole, itraconazole, posaconazole, artesunate-pyronaridine, ritonavir, indinavir, nelfinavir, atazanavir, glecaprevir-pibrentasvir, simeprevir, ledipasvir-sofosbuvir, verapamil, diltiazem, dronedarone, propafenone, quinidine, cyclosporine, valspodar, or milk thistle [Silybum marianum])
* Use of aldosterone antagonist (eg, spironolactone, eplerenone) and phenytoin within 4 weeks before the start of the study intervention

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1310 (Estimated)
Dates: Start 2023-12-31 (Actual); Primary Completion 2028-08-02 (Estimated); Study Completion 2028-08-02 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) in Androgen Receptor Ligand Binding Domain (AR LBD) Mutation-Positive Participants | Up to ~54 months
  OS is defined as time from randomization to death due to any cause. OS in AR LBD mutation-positive participants will be reported for each study arm.
OS in AR LBD Mutation-Negative Participants | Up to ~54 months
  OS is defined as time from randomization to death due to any cause. OS in AR LBD mutation-negative participants will be reported for each study arm.

SECONDARY OUTCOMES:
Radiographic Progression-free Survival (rPFS) Per Prostate Cancer Working Group-modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review in AR LBD Mutation-Positive Participants | Up to ~36 months
  rPFS is defined as the time from randomization to the first documented disease progression per Prostate Cancer Working Group (PCWG)-modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by Blinded Independent Central Review (BICR) or death due to any cause, whichever occurs first. rPFS in AR LBD mutation-positive participants will be reported for each study arm.
rPFS Per Prostate Cancer Working Group-modifiedRECIST 1.1 as Assessed by Blinded Independent Central Review in AR LBD Mutation-Negative Participants | Up to ~36 months
  rPFS is defined as the time from randomization to the first documented disease progression per Prostate Cancer Working Group (PCWG)-modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by Blinded Independent Central Review (BICR) or death due to any cause, whichever occurs first. rPFS in AR LBD mutation-positive participants will be reported for each study arm.
Time to Initiation of the First Subsequent Anti-Cancer Therapy or Death (TFST) | Up to ~54 months
  TFST is defined as the time from randomization to initiation of the first subsequent anticancer therapy or death, whichever occurs first.
Objective Response (OR) | Up to ~54 months
  OR is determined by PCWG-modified RECIST 1.1 as assessed by BICR.
Duration of Response (DOR) | Up to ~54 months
  DOR is determined by PCWG-modified RECIST 1.1 as assessed by BICR.
Time to Pain Progression (TTPP) | Up to ~54 months
  TTPP is assessed by Brief Pain Inventory-Short Form (BPI-SF) Item 3 ("Worst Pain in 24 Hours") and opiate analgesic use (Analgesic Quantification Algorithm [AQA] Score).
Time to Prostate-specific Antigen (PSA) Progression | Up to ~54 months
  The time from randomization to PSA progression. The PSA progression date is defined as the date of either: 1) ≥25% increase and ≥2 ng/mL above the nadir, confirmed by a second value ≥3 weeks later if there is PSA decline from baseline 2) ≥25% increase and ≥2 ng/mL increase from baseline beyond 12 weeks if there is no PSA decline from baseline.
Time to First Symptomatic Skeletal-related Event (SSRE) | Up to ~54 months
  The time from randomization to the first occurrence of any of the following symptomatic skeletal-related events: 1) Use of EBRT to prevent or relieve skeletal symptoms; 2) new symptomatic pathologic bone fracture (vertebral or nonvertebral); 3) spinal cord compression; or 4) tumor-related orthopedic surgical intervention.
Number of Participants Who Experience an Adverse Event | Up to ~54 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants Who Discontinue Study Treatment Due to an Adverse Event | Up to ~54 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (281):
- United States (44):
  - University of California, Irvine (UCI) Health - UC Irvine Medical Center ( Site 0040), Orange, California
  - Stanford Cancer Center ( Site 0036), Palo Alto, California
  - Kaiser Permanente Riverside Medical Center ( Site 0099), Riverside, California
  - Anschutz Cancer Pavilion ( Site 0046), Aurora, Colorado
  - University of Colorado Health - Highlands Ranch Hospital ( Site 0111), Highlands Ranch, Colorado
  - Colorado Clinical Research ( Site 0067), Lakewood, Colorado
  - University of Colorado Health - Lone Tree Medical Center ( Site 0112), Lone Tree, Colorado
  - Yale-New Haven Hospital-Yale Cancer Center ( Site 0064), New Haven, Connecticut
  - Florida Cancer Specialists - South ( Site 7003), Fort Myers, Florida
  - Bruce W. Carter Veterans Affairs Medical Center ( Site 0082), Miami, Florida
  - University of Miami Hospital and Clinics, Sylvester Cancer Center ( Site 0051), Miami, Florida
  - University of Illinois at Chicago ( Site 0105), Chicago, Illinois
  - University of Chicago Medical Center ( Site 0045), Chicago, Illinois
  - University of Iowa ( Site 0047), Iowa City, Iowa
  - University of Kentucky Chandler Medical Center ( Site 0048), Lexington, Kentucky
  - Ochsner Clinic Foundation ( Site 0108), New Orleans, Louisiana
  - Baltimore Veterans Affairs Medical Center ( Site 0069), Baltimore, Maryland
  - Greenebaum Comprehensive Cancer Center ( Site 0049), Baltimore, Maryland
  - Henry Ford Hospital ( Site 0015), Detroit, Michigan
  - M Health Fairview Clinics and Surgery Center ( Site 0019), Minneapolis, Minnesota
  - Metro-Minnesota Community Clinical Oncology ( Site 0014), Saint Louis Park, Minnesota
  - Washington University School of Medicine-Internal Medicine/Oncology ( Site 0062), St Louis, Missouri
  - University Of Nebraska Medical Center-Oncology/Hematology ( Site 0095), Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada ( Site 0010), Las Vegas, Nevada
  - Atlantic Health System Morristown Medical Center ( Site 0115), Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey ( Site 0033), New Brunswick, New Jersey
  - James J. Peters VA Medical Center ( Site 0088), The Bronx, New York
  - University Hospitals Cleveland Medical Center ( Site 0043), Cleveland, Ohio
  - Oregon Health and Science University ( Site 0028), Portland, Oregon
  - VA Portland Health Care System ( Site 0058), Portland, Oregon
  - AHN Allegheny General Hospital ( Site 0001), Pittsburgh, Pennsylvania
  - Ralph H. Johnson VA Health Care System (RHJVAHCS)-Urology ( Site 0083), Charleston, South Carolina
  - Avera Cancer Institute - Pierre ( Site 0118), Pierre, South Dakota
  - Avera Cancer Institute- Research ( Site 0094), Sioux Falls, South Dakota
  - Avera Cancer Institute - Yankton ( Site 0117), Yankton, South Dakota
  - SCRI Oncology Partners ( Site 7000), Nashville, Tennessee
  - Texas Oncology - Central/South Texas ( Site 8003), Austin, Texas
  - Texas Oncology - DFW ( Site 8001), Dallas, Texas
  - Texas Oncology - Gulf Coast ( Site 8002), The Woodlands, Texas
  - University of Virginia Health System ( Site 0054), Charlottesville, Virginia
  - VCU Health Adult Outpatient Pavillion ( Site 0061), Richmond, Virginia
  - Blue Ridge Cancer Care ( Site 0004), Roanoke, Virginia
  - Fred Hutchinson Cancer Center ( Site 0013), Seattle, Washington
  - MEDICAL COLLEGE OF WISCONSIN ( Site 0020), Milwaukee, Wisconsin
- Argentina (7):
  - Hospital Británico de Buenos Aires-Oncology ( Site 0202), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 0201), Mar del Plata, Buenos Aires
  - Instituto Alexander Fleming-Alexander Fleming ( Site 0206), Buenos Aires, Buenos Aires F.D.
  - Asociación de Beneficencia Hospital Sirio Libanés ( Site 0205), Buenos Aires, Buenos Aires F.D.
  - Sanatorio Parque ( Site 0208), Rosario, Santa Fe Province
  - Hospital Aleman-Oncology ( Site 0207), Buenos Aires
  - Fundacion Centro Oncologico de Integración Regional-Medical Oncology ( Site 0204), Mendoza
- Australia (5):
  - Dubbo Hospital ( Site 0235), Dubbo, New South Wales
  - Macquarie University-MQ Health Clinical Trials Unit ( Site 0234), Macquarie University, New South Wales
  - Westmead Hospital ( Site 0232), Westmead, New South Wales
  - Princess Alexandra Hospital-Cancer Care Serices ( Site 0237), Brisbane, Queensland
  - Peter MacCallum Cancer Centre-Parkville Cancer Clinical Trials Unit (PCCTU) ( Site 0230), Melbourne, Victoria
- Austria (3):
  - Medizinische Universität Graz-Innere Medizin Klin. Abt. Onkologie ( Site 0280), Graz, Styria
  - Ordensklinikum Linz GmbH Elisabethinen-Urologie ( Site 0276), Linz, Upper Austria
  - Klinikum Wels-Grieskirchen GmbH ( Site 0279), Wels, Upper Austria
- Brazil (8):
  - Hospital Santa Rita de Cassia-Centro de Pesquisa Clínica ( Site 0320), Vitória, Espírito Santo
  - Obras Sociais Irma Dulce ( Site 0302), Salvador, Estado de Bahia
  - Hospital Felicio Rocho ( Site 0317), Belo Horizonte, Minas Gerais
  - Hospital Mario Penna ( Site 0309), Belo Horizonte, Minas Gerais
  - Hospital Universitário Evangélico Mackenzie-Centro de Oncologia Mackenzie ( Site 0314), Curitiba, Paraná
  - Clínica de Neoplasias Litoral ( Site 0305), Itajaí, Santa Catarina
  - Hospital Universitário São Francisco de Assis - Bragança Paulista ( Site 0308), Bragança Paulista, São Paulo
  - A. C. Camargo Cancer Center ( Site 0310), São Paulo, São Paulo
- Canada (8):
  - Cross Cancer Institute ( Site 0332), Edmonton, Alberta
  - The Ottawa Hospital - General Campus-The Ottawa Hospital Cancer Centre ( Site 0336), Ottawa, Ontario
  - Sunnybrook Research Institute ( Site 0331), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 0330), Toronto, Ontario
  - Centre Intégré de Santé et de Services Sociaux de la Montérégie-Centre ( Site 0328), Greenfield Park, Quebec
  - Centre Hospitalier de l'Université de Montréal ( Site 0326), Montreal, Quebec
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus ( Site 0327), Québec, Quebec
  - Centre intégré universitaire de santé et de services sociaux de l'Estrie - Centre Hospitalier Univer ( Site 0329), Sherbrooke, Quebec
- Chile (7):
  - IC La Serena Research ( Site 0356), La Serena, Coquimbo Region
  - Clinical Research Chile SpA ( Site 0358), Valdivia, Los Ríos Region
  - Clinica Universidad Catolica del Maule-Oncology ( Site 0355), Talca, Maule Region
  - FALP ( Site 0353), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile-Hemato-Oncology ( Site 0354), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 0351), Santiago, Region M. de Santiago
  - Bradford Hill Norte ( Site 0357), Antofagasta
- China (39):
  - Second Affiliated hospital of Anhui Medical University-Urology ( Site 0408), Hefei, Anhui
  - Peking University First Hospital-Urology ( Site 0390), Beijing, Beijing Municipality
  - Beijing Friendship Hospital Affiliate of Capital University ( Site 0396), Beijing, Beijing Municipality
  - Beijing Cancer hospital-Urinary Surgery ( Site 0395), Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University ( Site 0427), Chongqing, Chongqing Municipality
  - Chongqing University Cancer Hospital ( Site 0416), Chongqing, Chongqing Municipality
  - Southwest Hospital of Third Military Medical University ( Site 0420), Chongqing, Chongqing Municipality
  - Chongqing Three Gorges Central Hospital's ( Site 0426), Chongqing, Chongqing Municipality
  - The First Affiliated Hospital Of Fujian Medical University-Urology ( Site 0414), Fuzhou, Fujian
  - The First Affiliated hospital of Xiamen University-Urology ( Site 0415), Xiamen, Fujian
  - The First Affiliated Hospital of Guangzhou Medical University ( Site 0412), Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center-Internal medicine ( Site 0413), Guangzhou, Guangdong
  - Tongji Hospital Tongji Medical,Science & Technology ( Site 0407), Wuhan, Hubei
  - Hubei Cancer Hospital-Urinary surgery ( Site 0406), Wuhan, Hubei
  - Hunan Cancer Hospital ( Site 0405), Changsha, Hunan
  - First Huai'an Hospital Affiliated to Nanjing Medical University ( Site 0436), Huaian, Jiangsu
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School-Urology ( Site 0377), Nanjing, Jiangsu
  - Affiliated hospital of Jiangnan university ( Site 0434), Wuxi, Jiangsu
  - Jiangxi Cancer Hospital ( Site 0386), Nanchang, Jiangxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University ( Site 0394), Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University-Oncology ( Site 0393), Xi'an, Shaanxi
  - Yantai Yuhuangding Hospital ( Site 0397), Yantai, Shandong
  - Zhongshan Hospital of Fudan University (0430), Shanghai, Shangai
  - Fudan University Shanghai Cancer Center-Urology department ( Site 0376), Shanghai, Shanghai Municipality
  - Huadong Hospital Affiliated to Fudan University-Urology ( Site 0388), Shanghai, Shanghai Municipality
  - The Third People's Hospital of Chengdu (CDTPH) ( Site 0428), Chengdu, Sichuan
  - West China Hospital, Sichuan University-Urology Surgery ( Site 0417), Chengdu, Sichuan
  - Nanchong Central Hospital-urology ( Site 0422), Nanchong, Sichuan
  - Suining Central Hospital ( Site 0437), Suining, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital ( Site 0392), Tianjin, Tianjin Municipality
  - The Second Hospital of Tianjin Medical University ( Site 0391), Tianjin, Tianjin Municipality
  - Xinjiang Medical University Cancer Hospital - Urumqi-Urology ( Site 0419), Ürümqi, Xinjiang
  - The Second Affiliated Hospital Of Kunming Medical University ( Site 0429), Kunming, Yunnan
  - Yunnan Province Cancer Hospital ( Site 0418), Kunming, Yunnan
  - Zhejiang Provincial People's Hospital-Urology ( Site 0378), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 0435), Hangzhou, Zhejiang
  - The First Hospital of Jiaxing-urology ( Site 0380), Jiaxing, Zhejiang
  - The First Affiliated Hospital of Ningbo University ( Site 0383), Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University-Urology Surgery ( Site 0379), Wenzhou, Zhejiang
- Colombia (6):
  - Clinica Colsanitas S.A, Sede Clínica Universitaria Colombia-Center Investigator ( Site 0501), Bogotá, Bogota D.C.
  - Sociedad De Oncología y Hematología Del Cesar SAS-Oncology ( Site 0502), Valledupar, Cesar Department
  - IMAT S.A.S ( Site 0504), Montería, Departamento de Córdoba
  - Fundación Cardiovascular de Colombia ( Site 0503), Piedecuesta, Santander Department
  - Fundación Valle del Lili ( Site 0505), Cali, Valle del Cauca Department
  - Clínica Imbanaco S.A.S ( Site 0509), Cali, Valle del Cauca Department
- Czechia (4):
  - Masarykuv onkologicky ustav-Klinika komplexni onkologicke pece ( Site 0553), Brno, Brno-mesto
  - Fakultni nemocnice Ostrava-Klinika onkologicka ( Site 0554), Ostrava, Moravskoslezský kraj
  - Fakultni nemocnice Olomouc-Onkologicka klinika ( Site 0555), Olomouc, Olomoucký kraj
  - Fakultni nemocnice v Motole-Onkologicka klinika 2. LF UK a FN Motol ( Site 0551), Prague, Praha 5
- Denmark (3):
  - Rigshospitalet ( Site 0576), Copenhagen, Capital Region
  - Odense Universitetshospital-Department of oncology ( Site 0579), Odense, Region Syddanmark
  - Vejle Sygehus ( Site 0578), Vejle, Region Syddanmark
- Finland (3):
  - Kuopion Yliopistollinen Sairaala ( Site 0603), Kuopio, Northern Savonia
  - Tampereen yliopistollinen sairaala ( Site 0604), Tampere, Pirkanmaa
  - Turku University Hospital-Department of Oncology ( Site 0601), Turku, Southwest Finland
- France (7):
  - Institut de cancérologie Strasbourg Europe (ICANS) ( Site 0627), Strasbourg, Alsace
  - Centre Hospitalier Universitaire de Nîmes - Institut de Cancérologie du Gard - Hôpital Universitaire ( Site 0630), Nîmes, Gard
  - Centre Eugène Marquis Rennes - Centre de Lutte Contre le Cancer ( Site 0632), Rennes, Ille-et-Vilaine
  - Centre Jean Perrin - Centre Régional de Lutte contre le Cancer d'Auvergne ( Site 0629), Clermont-Ferrand, Puy-de-Dome
  - Centre Hospitalier de la Côte Basque ( Site 0633), Bayonne, Pyrenees-Atlantiques
  - Gustave Roussy ( Site 0626), Villejuif, Val-de-Marne
  - Hôpital Européen Georges Pompidou ( Site 0628), Paris
- Germany (8):
  - klinikum rechts der isar der technischen universität münchen-Urologische Klinik und Poliklinik ( Site 0696), Munich, Bavaria
  - HELIOS Kliniken Schwerin ( Site 0694), Schwerin, Mecklenburg-Vorpommern
  - Universitätsklinikum Bonn-Klinik und Poliklinik für Urologie und Kinderurologie ( Site 0680), Bonn, North Rhine-Westphalia
  - Universitätsklinikum Münster - Albert Schweitzer Campus-Klinik für Urologie ( Site 0678), Münster, North Rhine-Westphalia
  - Universitätsklinikum Schleswig-Holstein-Klinik für Urologie ( Site 0691), Lübeck, Schleswig-Holstein
  - Universitätsklinikum Jena-Klinik und Poliklinik für Urologie ( Site 0682), Jena, Thuringia
  - Charité Universitaetsmedizin Berlin - Campus Mitte ( Site 0679), Berlin
  - Universitaetsklinikum Hamburg-Eppendorf-Onkologisches Zentrum ( Site 0705), Hamburg
- Hong Kong (2):
  - Queen Mary Hospital ( Site 0727), Hong Kong
  - Prince of Wales Hospital ( Site 0730), Shatin
- Hungary (4):
  - Bacs-Kiskun Varmegyei Oktatokorhaz-Onkoradiologiai Kozpont ( Site 0752), Kecskemét, Bács-Kiskun county
  - Nograd Varmegyei Szent Lazar Korhaz-Onkologia es Sugarterapias Osztaly ( Site 0761), Salgótarján, Nógrád megye
  - Országos Onkológiai Intézet-Urogenitális Tumorok és Klinikai Farmakológiai Osztály ( Site 0756), Budapest, Pest County
  - Debreceni Egyetem Klinikai Kozpont-Onkológiai Klinika ( Site 0758), Debrecen
- Ireland (2):
  - St. Vincent's University Hospital ( Site 0802), Dublin, Dublin
  - Tallaght University Hospital ( Site 0801), Dublin
- Israel (6):
  - Emek Medical Center ( Site 0830), Afula
  - Rambam Health Care Campus-Oncology Division ( Site 0826), Haifa
  - Hadassah Medical Center ( Site 0833), Jerusalem
  - Meir Medical Center. ( Site 0832), Kfar Saba
  - Rabin Medical Center ( Site 0828), Petah Tikva
  - Sheba Medical Center ( Site 0827), Ramat Gan
- Italy (3):
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori"-Oncologia Medica ( Site 0879), Meldola, Emilia-Romagna
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 0877), Milan, Lombardy
  - Ospedale San Raffaele-Oncologia Medica ( Site 0876), Milan
- Japan (30):
  - Toho University Sakura Medical Center ( Site 0906), Sakura, Chiba
  - Ehime University Hospital ( Site 0918), Tōon, Ehime
  - Hospital of the University of Occupational and Environmental Health, Japan ( Site 0921), Kitakyushu, Fukuoka
  - Kurume University Hospital ( Site 0920), Kurume, Fukuoka
  - Asahikawa Medical University Hospital ( Site 0901), Asahikawa, Hokkaido
  - Sapporo Medical University Hospital ( Site 0902), Sapporo, Hokkaido
  - Hokkaido University Hospital ( Site 0931), Sapporo, Hokkaido
  - Kobe University Hospital ( Site 0914), Kobe, Hyōgo
  - Kanazawa Medical University Hospital ( Site 0909), Mukai-awagasaki, Ishikawa-ken
  - Kagawa University Hospital ( Site 0917), Kita, Kagawa-ken
  - Yokohama City University Medical Center ( Site 0908), Yokohama, Kanagawa
  - National Hospital Organization Nagasaki Medical Center ( Site 0923), Ōmura, Nagasaki
  - Nara Medical University Hospital ( Site 0915), Kashihara, Nara
  - Nanbu Tokushukai Hospital ( Site 0930), Shimajiri, Okinawa
  - Kansai Medical University Hospital ( Site 0912), Hirakata, Osaka
  - Bell Land General Hospital ( Site 0913), Sakai, Osaka
  - The University of Osaka Hospital ( Site 0911), Suita, Osaka
  - Saga-Ken Medical Centre Koseikan ( Site 0922), Saga, Saga-ken
  - The Jikei University Hospital ( Site 0907), Minato, Tokyo
  - Akita University Hospital ( Site 0904), Akita
  - Kyushu University Hospital ( Site 0919), Fukuoka
  - Fukushima Medical University Hospital ( Site 0933), Fukushima
  - Gifu University Hospital ( Site 0910), Gifu
  - Hiroshima University Hospital ( Site 0916), Hiroshima
  - Kagoshima University Hospital ( Site 0929), Kagoshima
  - National Hospital Organization Kumamoto Medical Center ( Site 0924), Kumamoto
  - Miyazaki Prefectural Miyazaki Hospital ( Site 0927), Miyazaki
  - University of Miyazaki Hospital ( Site 0926), Miyazaki
  - Nagano Municipal Hospital ( Site 0932), Nagano
  - National Hospital Organization Oita Medical Center ( Site 0925), Ōita
- Malaysia (5):
  - Hospital Sultan Ismail ( Site 1081), Johor Bahru, Johor
  - University Malaya Medical Centre ( Site 1077), Lembah Pantai, Kuala Lumpur
  - National Cancer Institute ( Site 1079), Putrajaya, Putrajaya
  - Sarawak General Hospital-Radiotherapy Unit ( Site 1076), Kuching, Sarawak
  - Hospital Kuala Lumpur-Radiotherapy and Oncology ( Site 1078), Kuala Lumpur
- Mexico (5):
  - CIO - Centro de Inmuno-Oncología de Occidente ( Site 1103), Guadalajara, Jalisco
  - Quemex Medical and Research ( Site 1112), Mexico City, Mexico City
  - Filios Alta Medicina ( Site 1106), Monterrey, Nuevo León
  - Medical Care and Research SA de CV ( Site 1108), Mérida, Yucatán
  - Centro de Investigacion Clinica de Oaxaca ( Site 1109), Oaxaca City
- Netherlands (11):
  - Radboudumc-Medical Oncology ( Site 1152), Nijmegen, Gelderland
  - Zuyderland Medical Centre-Trialbureau Interne Geneeskunde ( Site 1163), Sittard-Geleen, Limburg
  - VieCuri Medisch Centrum ( Site 1173), Venlo, Limburg
  - ETZ Elisabeth-Internal Medicine ( Site 1160), Tilburg, North Brabant
  - Nederlands Kanker Instituut - Antoni van Leeuwenhoek - NKI-AVL ( Site 1153), Amsterdam, North Holland
  - Amsterdam UMC, locatie VUmc ( Site 1156), Amsterdam, North Holland
  - Spaarne Gasthuis - Hoofddorp-Oncology ( Site 1170), Hoofddorp, North Holland
  - Medische Centrum Leeuwarden ( Site 1172), Leeuwarden, Provincie Friesland
  - Franciscus Gasthuis & Vlietland, Locatie Vlietland ( Site 1151), Schiedam, South Holland
  - Haga Ziekenhuis locatie Leyweg-Oncology ( Site 1164), The Hague, South Holland
  - Meander Medisch Centrum ( Site 1157), Amersfoort, Utrecht
- New Zealand (2):
  - Tauranga Hospital-Bay of Plenty Clinical Trials Unit ( Site 1201), Tauranga, Bay of Plenty
  - Dunedin Hospital-Southern Blood and Cancers Service ( Site 1203), Dunedin, Otago
- Norway (3):
  - Akershus Universitetssykehus-Onkologisk avdeling ( Site 1227), Lørenskog, Akershus
  - St. Olavs Hospital-Kreftklinikken ( Site 1231), Trondheim, Sor-Trondelag
  - Sykehuset Østfold Kalnes ( Site 1228), Sarpsborg, Østfold fylke
- Peru (6):
  - Instituto Regional de Enfermedades Neoplasicas del Centro (IREN CENTRO) ( Site 1258), Concepción, Departamento de Junín
  - Clínica Sánchez Ferrer ( Site 1261), Trujillo, La Libertad
  - Aliada-Oncologìa ( Site 1257), Lima
  - IPOR Instituto Peruano de Oncología & Radioterapia-Centro de Investigación ( Site 1254), Lima
  - Oncosalud-Clinical Research ( Site 1260), Lima
  - INSTITUTO NACIONAL DE ENFERMEDADES NEOPLASICAS-Medical Oncology ( Site 1256), Lima
- Poland (7):
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka-Ambulatorium Chemioterapii ( Site 1302), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Regionalny Szpital Specjalistyczny im. dr. Władyslawa Biegańskiego ( Site 1316), Grudziądz, Kuyavian-Pomeranian Voivodeship
  - Wojewodzki Szpital Zespolony im Ludwika Rydygiera w Toruniu ( Site 1304), Torun, Kuyavian-Pomeranian Voivodeship
  - Mazowiecki Szpital Wojewódzki w Siedlcach-Siedleckie Centrum Onkologii ( Site 1310), Siedlce, Masovian Voivodeship
  - Szpital Wojewódzki im. Mikoaja Kopernika w Koszalinie-Oddzial Dzienny Chemioterapii ( Site 1303), Koszalin, West Pomeranian Voivodeship
  - Zachodniopomorskie Centrum Onkologii ( Site 1311), Szczecin, West Pomeranian Voivodeship
  - Swietokrzyskie Centrum Onkologii, Samodzielny Publiczny Zakl-Klinika Onkologii Klinicznej, Dzial Ch ( Site 1318), Kielce, Świętokrzyskie Voivodeship
- Puerto Rico (3):
  - Puerto Rico Medical Research Center LLC ( Site 1354), Hato Rey
  - Ad-Vance Medical Research-Research ( Site 1353), Ponce
  - Pan American Center for Oncology Trials - Ciudadela ( Site 1351), San Juan
- Singapore (3):
  - National University Hospital ( Site 1376), Singapore, Central Singapore
  - National Cancer Centre Singapore ( Site 1377), Singapore, Central Singapore
  - Tan Tock Seng Hospital-Medical Oncology ( Site 1378), Singapore, Central Singapore
- South Korea (4):
  - Asan Medical Center-Oncology ( Site 1402), Songpagu, Seoul
  - Seoul National University Hospital-Oncology ( Site 1401), Seoul
  - Severance Hospital, Yonsei University Health System-Medical oncology ( Site 1404), Seoul
  - Samsung Medical Center ( Site 1405), Seoul
- Spain (7):
  - Hospital Jerez de la Frontera ( Site 1427), Jerez de la Frontera, Cadiz
  - Hospital Universitario Ramón y Cajal-Medical Oncology ( Site 1431), Madrid, Madrid, Comunidad de
  - Hospital Universitario 12 de Octubre-Medical Oncology ( Site 1433), Madrid, Madrid, Comunidad de
  - Complexo Hospitalario Universitario de Ourense ( Site 1426), Ourense, Orense
  - Fundación Instituto Valenciano de Oncología-Oncologico ( Site 1430), Valencia, Valenciana, Comunitat
  - Hospital Lucus Augusti-Oncology ( Site 1432), Lugo
  - HOSPITAL UNIVERSITARIO VIRGEN DEL ROCIO-Medical Oncology ( Site 1428), Seville
- Sweden (3):
  - Karolinska Universitetssjukhuset Solna ( Site 1478), Stockholm, Stockholm County
  - Akademiska sjukhuset-Blod- och tumörsjukdomar ( Site 1477), Uppsala, Uppsala County
  - Sahlgrenska Universitetssjukhuset ( Site 1479), Gothenburg, Västra Götaland County
- Taiwan (5):
  - China Medical University Hospital-Department of Urology ( Site 1503), Taichung
  - National Cheng Kung University Hospital-Urology ( Site 1502), Tainan
  - National Taiwan University Hospital-Urology ( Site 1506), Taipei
  - Taipei Veterans General Hospital ( Site 1505), Taipei
  - Chang Gung Medical Foundation-Linkou Branch-Medical Oncology ( Site 1504), Taoyuan District
- Thailand (4):
  - Chulalongkorn University ( Site 1530), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital ( Site 1531), Bangkok, Bangkok
  - Faculty of Medicine - Khon Kaen University ( Site 1526), Muang, Changwat Khon Kaen
  - Songklanagarind hospital ( Site 1527), Hat Yai, Changwat Songkhla
- Turkey (Türkiye) (8):
  - Baskent University Dr. Turgut Noyan Research and Training Center-ONCOLOGY ( Site 1554), Adana
  - Gulhane Egitim Arastirma Hastanesi ( Site 1558), Ankara
  - Hacettepe Universite Hastaneleri-oncology hospital ( Site 1551), Ankara
  - Memorial Ankara Hastanesi-Medical Oncology ( Site 1557), Ankara
  - Ankara Bilkent Şehir Hastanesi-Medical Oncology ( Site 1552), Ankara
  - Istanbul Universitesi Cerrahpasa-Medical Oncology ( Site 1555), Istanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 1553), Istanbul
  - Samsun Medical Park Hastanesi-medical oncology (1560), Samsun
- United Kingdom (6):
  - Addenbrooke's Hospital ( Site 1605), Cambridge, Cambridgeshire
  - The Royal Cornwall Hospital ( Site 1610), Truro, England
  - The Beatson West of Scotland Cancer Centre ( Site 1603), Glasgow, Glasgow City
  - Charing Cross Hospital-Oncology Research ( Site 1606), London, Hammersmith and Fulham
  - University College London Hospital ( Site 1612), London, London, City of
  - The Christie NHS Foundation Trust ( Site 1608), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/